CLINICAL TRIAL: NCT00399282
Title: Comparison of the Effects of Simultaneous Administration of Vitamin E and Omega-3 Fatty Acids in Patients With Rheumatoid Arthritis
Brief Title: Omega-3 and Vitamin E Supplementation in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NNFTRI-2484
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Health related quality of life; Omega 3 fatty acids; Vitamin E
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Omega-3 and Vitamin E supplementation

SUMMARY:
The purpose of this study is to determine whether simultaneous supplementation with omega-3 fatty acids and vitamin E is effective in the treatment of patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether simultaneous supplementation with omega-3 fatty acids and vitamin E is effective in the treatment of patients with rheumatoid arthritis.

Most of studies on omega-3 fatty acids (omega-3) supplementation in patients with rheumatoid arthritis (RA) have clearly shown potentially beneficial changes in cytokine and eicosanoid metabolism. The overall clinical improvement, however, has been only moderate. One explanation is that an increased intake of omega-3 leads to a reduction in the availability of antioxidants and an increased generation of lipid peroxides. The majority of the anti-inflammatory drugs routinely used nowadays are COX (cyclo-oxygenase) inhibitors. Mechanism of COX II inhibitors is similar of omega-3. So, it is difficult to differentiate omega-3 net effects in some situations. Existing clinical trials on omega-3 and vitamin E (Vit E) are sometimes questioned due to using omega-6 fatty acids as placebo and neglecting omega-6 fatty acid intake in the diet. A comprehensive randomized controlled double-blind trial would have omega-6 fatty acids served as placebo in patients who are well matched in terms of therapies and drugs.

Comparison(s): Comparison of groups supplemented with omega-3, omega-3 with Vit E, and placebo (Medium chain triglycerides: MCT).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of rheumatoid arthritis according American college of rheumatology (ACR)

Exclusion Criteria:

* Infection
* Major joint malformations
* Simultaneous diseases like metabolic and gastrointestinal
* Being class IV according to ACR
* Drug dose fluctuations
* History of Vit E and/or omega-3 supplements during past six months
* Gastric irrigations

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75
Dates: Start 2006-10; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Score on Persian version of health assessment questionnaire (PE-HAQ) at 0, 6 and 12 weeks
Disease activity score at 0, 6 and 12 weeks
Duration of morning stiffness (in minutes) at 0, 6 and 12 weeks
Joint pain intensity, on a five-point scale (0, absent) at 0, 6 and 12 weeks
Onset of fatigue (in minutes) after walking at 0, 6 and 12 weeks
Ritchie's articular index for pain joints at 0, 6 and 12 weeks
Right and left grip strength (in mmHg) measured with a sphygmomanometer cuff inflated to 20 mmHg at 0, 6 and 12 weeks
Patient's global assessment of disease activity (0 to 10 cm visual analog scale: 0, symptom free; 10, very severe) at 0, 6 and 12 weeks
Classification of functional status in RA according to revised criteria of the American
College of Rheumatology at 0, 6 and 12 weeks
Patient's satisfaction in activities of daily living based on a Persian version of Health Assessment Questionnaire (PE-HAQ) at 0, 6 and 12 weeks

SECONDARY OUTCOMES:
TNF-alpha at 0, 6 and 12 weeks
IL-1 beta at 0, 6 and 12 weeks
C-reactive protein at 0, 6 and 12 weeks
Erythrocyte sedimentation rate at 0, 6 and 12 weeks
Malondialdehyde at 0, 6 and 12 weeks
Systolic blood pressure at 0, 6 and 12 weeks
Diastolic blood pressure at 0, 6 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Reza Rastmanesh, Ph.D., Principal Investigator — National Nutrition and Food Sciences Technology Institute
Locations (1):
- Rheumatology Research Center (RRC), Tehran University for medical Sciences (TUMS), Tehran, Iran